CLINICAL TRIAL: NCT05572723
Title: Comparison of the Effects of Remifentanil and Dexmedetomidine Administered Under General Anesthesia in Rhinoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Zeynep Ersoy, Assistant professor, Baskent University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: KA 22/12
Record Dates: First submitted 2022-09-23; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Rhinoplasty; Dexmedetomidine; Remifentanil
Keywords: Remifentanil; dexmedetomidine; pain; recovery; shivering
MeSH Terms: conditions — Pain | interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Remifentanil (Active Comparator): Remifentanil group was initially to receive remifentanil (group R), 0.01-0.2 g/kg/min without intraoperative loading.
  Interventions: Drug: Remifentanil 2 MG
- Group Dexmedetomidine (Active Comparator): Dexmedetomidine group, dexmedetomidine (group D) was initiated with a bolus of 1 mg/kg and received 0.2-0.7 g/kg per hour as an infusion during surgery.
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: Remifentanil 2 MG — Remifentanil is an opioid; it has sedative, analgesic, and sympatholytic properties.
  Arms: Group Remifentanil
Drug: dexmedetomidine — Studies show that dexmedetomidine is superior to currently commonly used remifentanil in terms of intraoperative blood pressure control and postoperative pain.
  Dexmedetomidine, an alpha-2-adrenoceptor agonist, has sympatholytic, sedative, anesthetic, analgesic, and vasoconstrictor effects. It lowers blood pressure by decreasing plasma norepinephrine and epinephrine levels, thereby reducing intraoperative bleeding. Dexmedetomidine is defined as an analgesic that is now widely used to induce and maintain anesthesia and to control postoperative pain, and is defined as an analgesic that does not cause respiratory depression and neurocognitive impairment. Many studies have shown that the use of perioperative dexmedetomidine reduces the stress response to anesthetic induction and surgery and provides hemodynamic stability.
  Arms: Group Dexmedetomidine

SUMMARY:
The investigators compared the effects of remifentanil and dexmedetomidine administered under general anesthesia on hemodynamics, postoperative pain, recovery, postoperative nausea, vomiting, shivering, patient's and surgeon's satisfaction in patients undergoing elective rhinoplasty. A single-center, prospective, blinded, randomized controlled trial. After the approval of the hospital ethics committee (KA22/12), fifty volunteers aged 18-65 years who underwent rhinoplasty under elective conditions accepted the study in the American Society of Anesthesiologists (ASA) I-III class. The patients were randomly divided into the remifentanil group (group R) and the dexmedetomidine group (group D). Group R (n=25) was initially to receive remifentanil 0.01-0.2 g/kg/min without intraoperative loading. Group D (n=25) dexmedetomidine, was initiated with a bolus of 1 mg/kg and received 0.2-0.7 g/kg per hour as an infusion during surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients who will have rhinoplasty surgery American Society of Anesthesiologists (ASA) I- II class

Exclusion Criteria:

Patients with end-stage liver or kidney disease Uncontrolled hypertension Any type of atrioventricular block, pacemaker Heart failure Diabetes mellitus Chronic obstructive or interstitial lung disease, severe asthma Neurological or psychiatric disease, substance abuse Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | During surgery
  The investigators compare the stability of mean arterial pressure.
Postoperative pain | Up to 30 minutes after the patient wakes up.
  The investigators compare the effect of remifentanil and dexmedetomidine on postoperative pain. The patients pain level was assessed using the numeric pain scale (Between 0-10, 0 = no pain, 10 = worst pain).
Patient Recovery Time | Postoperative 1. hours
  The investigators compare the effect of remifentanil and dexmedetomidine on patient recovery time. The recovery time of the patient will be evaluated by calculating the time between extubated and discharged from the postoperative care unit.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting scores | postoperative first 6 hours and 24 hours
  The investigators compare the effect of remifentanil and dexmedetomidine on nausea and vomiting. The presence of PONV was assessed using the Verbal Descriptor Scale (Between 0-3, 0=no nausea, 1=mild, 2=moderate, 3=severe).
Patient satisfaction | Postoperative 6. hours
  The investigators will question patients' degree of postoperative satisfaction. The patient satisfaction scale was used to assess the surgical outcome (Between 1 - 5, 1 = very poor, 5 = very good).
Surgeon satisfaction | Postoperative 0. hours
  The investigators will question surgeons' degree of satisfaction. The surgical satisfaction scale was used to assess the surgical outcome (Between 1 - 5, 1 = very poor, 5 = excellent).

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Medical School, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No